CLINICAL TRIAL: NCT05882981
Title: Evaluation of Physical Performance of Young Adults With Increased Femoral Anteversion
Brief Title: Increased Femoral Anteversion and Physical Performance
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Assistant professor, Bezmialem Vakif University
Other Study IDs: DT-04
Record Dates: First submitted 2023-05-08; First posted 2023-05-31 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: High Femoral Anteversion; Muscle Strength; Flexibility; Functional Performance; Functional Capacity
MeSH Terms: interventions — 4-Acetamido-4'-isothiocyanatostilbene-2,2'-disulfonic Acid; Physical Functional Performance; Functional Residual Capacity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: 22 young adults aged 17-26 years with high femoral anteversion.
  Interventions: Other: Sit and reach test; Other: Hand grip strength measurement; Other: Back-leg-chest muscle strength measurement; Other: Functional performance; Other: Functional capacity
- Control group: 22 young adults aged 17-26 years with normal femoral anteversion
  Interventions: Other: Sit and reach test; Other: Hand grip strength measurement; Other: Back-leg-chest muscle strength measurement; Other: Functional performance; Other: Functional capacity

INTERVENTIONS:
Other: Sit and reach test — It will be used to measure the flexibility of the participants.
Other: Hand grip strength measurement — Grip strength will be evaluated with a hand dynamometer in the position recommended by the American Association of Hand Therapists.
Other: Back-leg-chest muscle strength measurement — An analog Back Leg-Chest dynamometer will be used to evaluate general muscle strength.
Other: Functional performance — Single-leg and double-leg horizontal jump test will be used to evaluate lower extremity functional performance. The tests will be carried out according to the Eurofit test battery (Council of Europe, 1988).
Other: Functional capacity — Functional capacity will be evaluated with six minute walk test according to the ATS criteria.

SUMMARY:
It is important to determine how high femoral anteversion, which is one of the lower extremity malalignments, affects physical performance and to what extent it affects the daily life of the individual. As far as we know, there is no study on this subject except for a study conducted by Staheli et al. in 1977. Therefore, the investigators planned to determine whether and to what extent high femoral anteversion has an effect on physical performance in healthy young adults.

DETAILED DESCRIPTION:
One of the factors associated with problems in the lower extremity is changes in the angle of femoral anteversion. High femoral anteversion causes pathological changes in the sagittal and coronal planes, especially in the transverse plane, and changes the gait biomechanics. Femoral anteversion angle; It is the angle formed by the plane of the femoral condyle and the plane passing through the femoral neck and the femoral head. The femoral anteversion angle, which is 55°-60° in the intrauterine period, is approximately 30° at birth. In the postnatal period, with normal growth, it decreases by 1.5° per year until the age of 15, decreasing to 26° at the age of 5, 21° at the age of 9 and 15° at the age of 16.

Toe-in gait pattern may be due to foot deformity (metatarsus adductus) and/or transverse alignment disorder of the long bones (tibial torsion and/or femoral anteversion height). When the angle of anterversion is high, walking with the feet turned in is 30.9% at the age of 4, 15% at the age of 4, and around 4% in adults. High femoral anteversion, which is the most common cause of inward walking in early childhood, is mostly seen symmetrically, with a higher incidence in girls and hypermobile children. Most cases are idiopathic and some patients have a familial predisposition.

Alignment disorders in the lower extremities can cause problems affecting other segments of the body, postural disorders and problems in the musculoskeletal system, as well as affect physical performance. The study, which will examine the physical performance status of young adults with high femoral anteversion, will be carried out as a cross-sectional study. The universe of the study will consist of students aged 17-26 who continue their education at the Faculty of Health Sciences of Bezmialem Vakıf University in the 2022-2023 academic year. Within the scope of our cross-sectional study, an application will be made for the approval of the Ethics Committee before the data are collected. The study, which will start after the permission is obtained, will be carried out in accordance with the Declaration of Helsinki. Evaluation and testing of all cases will be done at Bezmialem Vakif University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation. 22 subjects with high femoral anteversion angle and 22 subjects with normal femoral anteversion angle will be included in the study. Within the scope of the study, demographic information of all participants will be obtained with the evaluation form and clinical evaluations will be made. Flexibility with sit-reach test, hand grip strength with hydraulic hand dynamometer, general muscle strength with analog back-leg-chest dynamometer, functional performance with single-leg and double-leg horizontal jump tests, and functional capacities with 6-minute walking test will be evaluated. "Statistical Package for the Social Sciences (SPSS) 20.0 for Windows" package program will be used in the statistical analysis of the data obtained from the study which the investigators planned to evaluate physical performance in young adults with high femoral anteversion. All data will be analyzed with the Kolmogorov-Smirnov test to determine the distribution characteristics. In the study, descriptive statistics (mean±standard deviation, minimum-maximum, number and percentile) will be given for discrete and continuous variables. When the differences between two independent groups are evaluated, "t-Test in Independent Groups" in case the parametric test prerequisites are met; If not, the "Mann Whitney -U Test" will be used. "Chi-Square Test" will be used to determine the relationships between two discrete variables. When the variables meet the parametric test prerequisites, the correlation coefficients and statistical significance will be calculated with the "Pearson Test", when they do not, the correlation coefficients and statistical significance for the relations between the variables will be calculated with the "Spearman Test".

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral increased femoral anteversion
2. Hip internal rotation >60 degrees, external rotation <45
3. According to the Craig test, the anteversion angle is between 20-40 degrees
4. Absence of a history of neurological or psychiatric disease
5. Absence of intellectual disability to prevent participation in assessment and treatment
6. Not participating in any exercise/physiotherapy program in the last six months
7. Body mass index within normal limits (18.5-24.9 kg/m2)

Exclusion Criteria:

1. Having a history of BoNT-A or surgery in the last 6 months
2. Leg length inequality
3. Beighton score of 4 and above
4. Presence of 3rd degree pes planus

Ages: 17 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 22 young adults aged 17-26 years with high femoral anteversion.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Functional performance tests | One day
  Single-leg and double-leg horizontal jump test will be used to evaluate lower extremity functional performance. The tests will be carried out according to the Eurofit test battery (Council of Europe, 1988).
Functional capacity measurement | One day
  Functional capacity will be evaluated with six minute walk test according to the ATS criteria.

SECONDARY OUTCOMES:
Sit and reach test | One day
  It will be used to measure the flexibility of the participants.
Back-leg-chest muscle strength measurement | One day
  An analog Back Leg-Chest dynamometer will be used to evaluate general muscle strength.
Hand grip strength measurement | One day
  Grip strength will be evaluated with a hand dynamometer in the position recommended by the American Association of Hand Therapists.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided